CLINICAL TRIAL: NCT05039970
Title: A Real-World Study of the Effect of a Mobile Device-based Serious Health Game on Session Attendance in the National Diabetes Prevention Program
Brief Title: A Real-World Study of a Mobile Device-based Serious Health Game on Session Attendance in the National Diabetes Prevention Program
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: BioCentric, Inc. (Other)
Collaborators: Centers for Disease Control and Prevention (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 00055024
Record Dates: First submitted 2021-08-12; First posted 2021-09-10 (Actual); Last update posted 2022-11-02 (Actual); Status verified 2022-10

CONDITIONS: Diabetes Mellitus Risk; Diabetes Mellitus
Keywords: Prevention; Serious Health Game
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Intervention Model Description: This study will be a 2-arm parallel group cluster randomized, prospective, observational study in a real-world setting of organizations delivering the National DPP LCP. Cohorts will be randomized 1:1 to experimental or control arms. Participants in the experimental arm will download WellQuest™ and be instructed on use of the game. Participants in the control arm will proceed with routine National DPP participation. The study will focus on session attendance during the first 6 months of the 12-month program. Data will be received from 2 main sources. A secondary data analysis will be conducted on individual-level data collected by each participating organization (eg, demographics, sessions attended, body weight, minutes of physical activity). For the experimental arm only, individual-level data collected via the game use will include game downloads and daily time spent playing the game. Data on satisfaction will be collected via surveys disseminated through the game.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Arm - WellQuest™ Users (Experimental): Participants in National DPP groups randomized to the experimental arm will be instructed by lifestyle coaches to download the WellQuest™ game application and will receive instructions on how to use the game throughout the LCP.
  Interventions: Other: WellQuest™
- Control Arm (No Intervention): Participants in National DPP groups randomized to the control arm will proceed with their routine National DPP participation.

INTERVENTIONS:
Other: WellQuest™ — WellQuest™ is a mobile device-based serious health game.
  Arms: Experimental Arm - WellQuest™ Users

SUMMARY:
The overall prevalence of type 2 diabetes in the United States (US) is estimated at more than 30 million people, with an estimated 88 million more adults meeting the criteria for having prediabetes and being at risk for progressing to type 2 diabetes. The significant burden of diabetes, as well as the high individual and societal cost it bears, renders this disease among the highest public health priorities for the health authorities and policy makers. In response to the rising diabetes prevalence, the US Centers for Disease Control and Prevention (CDC) established the National Diabetes Prevention Program (National DPP) in 2010 as a framework for diabetes prevention by providing evidence-based, affordable, and high-quality lifestyle change programs (LCPs). The National DPP LCP is a yearlong education-based curriculum focused on achieving modest weight loss (5% to 7%) and increasing participants' physical activity to reduce the risk of progressing to type 2 diabetes. To ensure high-quality programs and meaningful impact on participants, the CDC sets standards for organizations that wish to offer an LCP through the Diabetes Prevention Recognition Program (DPRP). The DPRP plays a critical role in ensuring that organizations can effectively deliver the evidence-based lifestyle change program with quality and fidelity. To achieve recognition status, organizations must periodically provide evidence that they are following a CDC-approved curriculum and achieving meaningful results on session attendance, body weight change, and physical activity minutes.

A recent analysis of National DPP data has shown that the attrition rates in this program are substantial and that they differ by age and race. Moreover, the attrition rates were inversely associated with the program success, as reflected by the LCP outcomes, and, specifically, participants' weight and level of physical activity. In view of these findings, the CDC is undertaking an effort to increase participant retention in the National DPP.

The proposed study will evaluate the pilot use of a free-of-charge mobile device-based serious health game (WellQuest™) within the frame of the National DPP LCP. WellQuest™ was designed with the goals to improve participant engagement and retention in the LCP, to encourage adoption and maintenance of healthy lifestyle habits among LCP participants, and to reinforce knowledge of the LCP curriculum.

ELIGIBILITY:
Inclusion Criteria:

* Enrollment in a qualifying National DPP program
* Body mass index (BMI) ≥25 kg/m2 for non-Asians and ≥23 kg/m2 for Asians.
* Have prediabetes identified by either a blood test or a self-reported risk test or have a history of gestational diabetes mellitus (GDM).

Exclusion Criteria:

* Participants cannot have a previous diagnosis of type 1 or type 2 diabetes, prior to enrollment in a National DPP.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 550 (Actual)
Dates: Start 2021-09-07 (Actual); Primary Completion 2022-10-31 (Actual); Study Completion 2022-10-31 (Actual)

PRIMARY OUTCOMES:
Number of Sessions Attended | 6 Months
  The primary outcome of this study is the number of sessions attended during the first 6 months following enrollment in a National DPP.

SECONDARY OUTCOMES:
Retention in National DPP 4 months and 6 months after enrollment. | 6 Months
  This outcome would be retention reported in number of sessions at 4 months and 6 months after enrollment.
Game downloads among participants randomized to the experimental arm | 6 Months
  Proportion of participants who download the game
Daily time spent playing the serious health game in participants who downloaded the game. | Six Months
  Amount of time in minutes spent by participants playing the game
Participants' game rating/Net Promoter Score or questionnaire. | Six Months
  Likert scale rating of participants' satisfaction questionnaire (willingness to recommend to others)

OTHER OUTCOMES:
Completeness of health data collected by the game | 6 Months
  Proportion of participants reporting health data via game
Comparability of health data collected by the game and data reported by the organization | 6 Months
  Percentage of health data reported in game versus the cohort data reported to CDC
Body weight (and/or body mass index [BMI]) change over time | 6 Months
  Change in body weight measured in pounds over study duration
Correlation between any weight loss (and/or BMI decrease) and game use | 6 Months
  Change in body weight measured in pounds in proportion to game use measured in minutes
Correlation of >5% weight loss and game use | 6 Months
  Game use measured in minutes among those who achieved >5% weight loss
Correlation of increased physical activity and game use | 6 Months
  Change in physical activity measured in minutes in proportion to game use measured in minutes
Correlation between retention in National DPP 6 months after enrollment and the amount of time spent playing the serious health game during the first month after enrollment | 6 Months
  Number of sessions in proportion to duration of game play during the first month (measured in minutes)
Number of sessions attended in the experimental cohort among those who downloaded the game and those who did not download the game | 6 Months
  Number of sessions attended as reported by the CDC among those who did and did not download the game as measured by number of downloads
Fitness tracker integration with the game. | 6 Months
  Proportion of game players who link fitness tracker to the game as measured by in-game analytics

CONTACTS AND LOCATIONS:
Overall Officials: Kevin Jarvis, PharmD, Principal Investigator — BioCentric, Inc.
Locations (1):
- BioCentric, Inc., Collingswood, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Information about the WellQuest™ game — http://www.wellquestgame.com